CLINICAL TRIAL: NCT07100483
Title: Prospective, Randomized Trial Comparing Left Atrial Cox-Maze IV, Tampa 2 or Encompass Alone, Ablation in the Surgical Management of Atrial Fibrillation
Brief Title: Comparing Surgical Management Methods of Atrial Fibrillation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Charles Willekes, Section Chief Cardiothoracic surgery, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1012
Record Dates: First submitted 2025-07-11; First posted 2025-08-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: AFib; Ablation; Cox IV; Tampa 2; Encompass; Box Lesion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a single enter prospective, randomized trial to compare the outcomes, specifically the freedom from atrial fibrillation at one year, and possibly up to five years, of three different approaches (Cox-Maze IV, Tampa 2, Encompass) to the cardiac surgical management of atrial fibrillation. All patients undergoing an elective, cardiac surgical procedure with documented preoperative AF, either paroxysmal or persistent, with a planned surgical ablation are potential candidates.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cox-Maze IV (Active Comparator): Lesion created around the pulmonary vein ostia (openings). Lesion to posterior (back) of the mitral annulus (fibrous ring around the mitral valve leaflets). Lesion from the 'box' to the left atrial appendage. There is also one lesion on the outside of the heart at the coronary sinus (main vein draining the heart)- not shown in this picture due to being on the outside of the heart. The Left Atrial Appendage will also be either excluded or removed.
  Interventions: Procedure: Atrial Fibrillation Ablation
- Tampa 2 (Active Comparator): Lesion created around the pulmonary vein ostia (openings). Lesion from the 'box' to the left atrial appendage Lesion from the left atrial appendage to the anterior (front) of the mitral annulus (fibrous ring around the mitral valve leaflets). This lesion is done through the left atrial appendage. The Left Atrial Appendage will also be either excluded or removed.
  Interventions: Procedure: Atrial Fibrillation Ablation
- Encompass Alone (Active Comparator): Lesion created around the pulmonary vein ostia (openings). The Left Atrial Appendage will also be either excluded or removed.
  Interventions: Procedure: Atrial Fibrillation Ablation

INTERVENTIONS:
Procedure: Atrial Fibrillation Ablation — Ablation of the heart to reduce Afib Occurrence

SUMMARY:
Compare the efficacy of the left atrial Cox-Maze IV lesion set versus the Tampa 2 lesion set versus the EnCompass ablation alone, in the surgical treatment of atrial fibrillation at one year post-operatively.

DETAILED DESCRIPTION:
This is a single center prospective, randomized trial to compare the outcomes, specifically the freedom from atrial fibrillation at one year, and possibly up to five years, of three different approaches to the cardiac surgical management of atrial fibrillation.

Several strategies to accomplish surgical ablation are acceptable and have been shown retrospectively to be successful. The Cox-Maze bi-atrial, left and right atrial lesions, ablation (whether III or IV) remains the gold standard by which all surgical ablations are compared. Further refinement in ablation technology and research has further suggested there is no difference between a left atrial ablation alone or bi-atrial ablation lesion set. For left atrial ablation alone, existent therapeutic options, which all meet equivalent standard of care, include a left atrial Cox-Maze IV , a Tampa 2 lesion set or utilizing a "box lesion" alone. Currently, there are no randomized, clinical trials demonstrating better efficacy (freedom from atrial fibrillation post-operatively) of one ablation strategy over another in patients undergoing cardiac surgery.

The rationale for the study is to demonstrate whether one ablation technique is more efficacious in the surgical treatment of AF. Should one technique prove superior it may clarify the question of which ablation strategy to utilize and encourage surgeons to implement a consistent approach to surgical ablation.

To our knowledge this study would be the first prospective, randomized trial in the United States comparing surgical lesion sets in the concomitant management of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a history of preoperative atrial fibrillation, either paroxysmal or persistent, requiring concomitant surgical ablation who are scheduled to undergo cardiac surgical procedure(s) to be performed on cardiopulmonary bypass
* Utilizing sternotomy approach requiring cardiopulmonary bypass
* Male or Female subjects between age 18 to 85 years of age

Exclusion Criteria:

* LVEF < 25%
* LAVI > 59ml/m②
* Presence of Pacemaker/AICD
* History of VT/VF, WPW
* Re-operative cardiac surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2032-09-15 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation | 30 days and 1 year
  Freedom from atrial fibrillation at 30 days and one year

SECONDARY OUTCOMES:
Prescribed Antiarrhythmic and anticoagulant drugs | 7 days and 1 year
  Antiarrhythmic and anticoagulant drugs at 7days and one year post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charles Willekes, MD, Principal Investigator — Corewell Health
Locations (1):
- Corewell Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No